CLINICAL TRIAL: NCT06369051
Title: Supporting Self-employment in Working-age Stroke Survivors
Brief Title: Supporting Self-employment in Young Adults with Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Suzanne HS Lo, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: YSEmploy
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): A new intervention developed to assist stroke survivors in becoming self-employed by developing entrepreneurial skills. It consists of one home visit, three online individual sessions, and four online group sessions held once a week for eight weeks.
  Interventions: Other: Self-employment support intervention
- Control (No Intervention): Usual stroke care services

INTERVENTIONS:
Other: Self-employment support intervention — A new intervention developed to assist stroke survivors in becoming self-employed by developing entrepreneurial skills. It consists of one home visit, three online individual sessions, and four online group sessions held once a week for eight weeks.
  Arms: Intervention

SUMMARY:
This project will investigate the effects of an 8-week theory-driven online/hybrid Self-employment Skill Building Intervention on the rate of self-employment, self-efficacy, life satisfaction, and psychosocial outcomes among working-age stroke survivors.

DETAILED DESCRIPTION:
A 2-arm randomised controlled trial will be conducted. Individuals aged 18-65 years old, with a first-ever/recurrent ischaemic/haemorrhagic stroke, and unemployed for at least 6 months will be recruited. Eligible participants will be randomly assigned to receive usual care or a new intervention with usual care. The intervention is aimed at assisting survivors in becoming self-employed by developing entrepreneurial skills. Outcomes including self-employment rate, self-efficacy, life satisfaction, emotional well-being, and community reintegration at baseline, immediately and 3 months after completing the intervention. Semi-structured interviews will be conducted with participants to elicit feedback on SSI.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old at the time of recruitment
* been clinically diagnosed with a first-ever/recurrent ischaemic/haemorrhagic stroke
* a Montreal Cognitive Assessment score (MoCA) >2nd percentile
* a paid job (full-time/part-time) at the recent onset of stroke
* been unemployed (not in paid, full-time/part-time job) for ≥6 months at the time of recruitment
* able to communicate in Cantonese and read Traditional Chinese.

Exclusion Criteria:

* diagnosed with transient ischaemic attack
* cerebrovascular events due to tumour
* diagnosed with a mental condition for example depression or schizophrenia
* incomprehensible speech
* receiving or awaiting to receive vocational programmes
* self-employed at the time of recruitment or planning to retire

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-employment rate | Change from baseline level to three months after completion of the intervention
  Self-employment work is defined as the active production of goods and/or services on one's own or with a small group for personal gains, including income, and is not performed for wages by employers. Work done by housewives, students, and volunteers is not included. A minimum of 10 hours per week should be committed to the work (25% of full-time work).(2,3) The participant's response will be rated as "Yes" or "No".

SECONDARY OUTCOMES:
Self-efficacy | Change from baseline level to three months after completion of the intervention
  Participants' self-efficacy in coping with stressful life events will be assessed by the 10-item General Self-Efficacy Scale (GSES) (Chinese version). Each item is rated on a 4-point scale (1=not at all true to 4=exactly true).
Life satisfaction | Change from baseline level to three months after completion of the intervention
  Participants' satisfaction with life will be measured by the Satisfaction with Life Scale (Chinese version). It contains 5 items that ask participants to rate their agreement with each statement on a 7-point scale (1=strongly disagree to 7=strongly agree).
Emotional well-being | Change from baseline level to three months after completion of the intervention
  Participants' emotional well-being will be measured by the 14-item Hospital Anxiety and Depression Scale (Chinese version). It has 2 subscales (anxiety and depression), and participants will rate their mood in the previous week on a 4-point scale (0=no not at all to 3=yes definitely). Summation of relevant item scores yields the subscale score (total=0-21).
Community reintegration | Change from baseline level to three months after completion of the intervention
  The 11-item Reintegration to Normal Living Index (Chinese version) will be used to assess participants' level of community reintegration.(44) It has 8 domains (mobility, daily self-care and work/activities, roles in family, relationships with others, presentation of self to others, coping skills). Participants will rate how well each item describes their situation (1=a small extent to 5=a great extent). Summation produces a total score that is normalised to 100 (range 25-100).

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lo, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Non-government organisations, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No